CLINICAL TRIAL: NCT01608659
Title: An Observational Retrospective Study to Evaluate Treatment Patterns of Botulinum Toxin Type A
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTXC-10-001
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Facial Rhytides
MeSH Terms: interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- botulinum toxin Type A: Previous treatment with botulinum toxin Type A for treatment of facial lines
  Interventions: Drug: botulinum toxin Type A

INTERVENTIONS:
Drug: botulinum toxin Type A — Previous treatment with botulinum toxin Type A for treatment of facial lines
  Other Names: BOTOX®; Xeomin®

SUMMARY:
This is a retrospective chart review to evaluate treatment patterns of botulinum toxin Type A for the treatment of facial lines.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated for glabellar lines (hyperfunctional facial lines) with botulinum toxin Type A preparation
* Received 2 treatment cycles wtih botulinum toxin Type A (BOTOX®) prior to at least 1 treatment with botulinum toxin Type A (Xeomin®)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated for glabellar lines (hyperfunctional facial lines) with botulinum toxin Type A
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2011-06-17 (Actual); Study Completion 2011-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Buenos Aires, Argentina

REFERENCES:
- [Background] Banegas RA, Farache F, Rancati A, Chain M, Gallagher CJ, Chapman MA, Caulkins CA. The South American Glabellar Experience Study (SAGE): a multicenter retrospective analysis of real-world treatment patterns following the introduction of incobotulinumtoxinA in Argentina. Aesthet Surg J. 2013 Sep 1;33(7):1039-45. doi: 10.1177/1090820X13503475. Epub 2013 Aug 29. PMID 23990584

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this retrospective chart review study, subjects received botulinum toxin Type A (BOTOX®) in study-defined Treatment Periods 1 and 3, and botulinum toxin Type A (Xeomin®) in Treatment Period 2. Data were evaluated as available for each Treatment Period.
Period: Overall Study
Arm/Group | Botulinum Toxin Type A
Started | 110
Completed | 94
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 110
Age, Customized [Number; unit: Participants]
  ≥30 and <40 years | 5
  ≥40 and <50 years | 31
  ≥50 and <60 years | 33
  ≥60 years | 35
  Missing | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Total Dose Per Treatment Period
Description: Average total dose per treatment period was defined as total treatment dose plus total touch-up dose plus total follow-up dose.
Time Frame: 24 Months
Population: All subjects enrolled in the study who were evaluated for this data point. N equals the number of subjects evaluated in each treatment period.
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 34
Units
  Treatment Period 1 (BOTOX®) N=34 | 49.2 (12.77)
  Treatment Period 2 (Xeomin®) N=34 | 48.1 (15.18)
  Treatment Period 3 (BOTOX®) N=16 | 45.8 (4.68)

2. Secondary Outcome: Inter-Injection Interval Duration of Each Treatment Period
Description: Inter-injection interval duration of each treatment period. Duration is defined as the number of days of an injection cycle.
Time Frame: 24 Months
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 110
Days
  Treatment Period 1 (BOTOX®) N=110 | 180.3 (94.40) [58 to 623]
  Treatment Period 2 (Xeomin®) N=106 | 144.3 (113.55) [13 to 658]
  Treatment Period 3 (BOTOX®) N=76 | 176.9 (91.43) [98 to 639]

3. Secondary Outcome: Percent of Subjects Reporting Satisfaction With Treatment Effects
Description: Percent of subjects reporting satisfaction with treatment effects per chart notes.
Time Frame: 24 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Subjects
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 80
Percentage of Subjects
  Treatment Period 1 (BOTOX®) N=80 | 99.0 (6.68)
  Treatment Period 2 (Xeomin®) N=74 | 33.7 (39.29)
  Treatment Period 3 (BOTOX®) N=67 | 90.3 (17.56)

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.